CLINICAL TRIAL: NCT02851251
Title: Multicenter Neonatal Eye Disease Screening in China
Status: Completed | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Peiquan Zhao, Professor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XH-16-019
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Eye Disease
Keywords: eye disease; neonatal eye disease; newborn; screening; multicenter
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
These exams are vital to protect healthy neonates from blindness. The purpose of this study is to better screen ocular disease in otherwise healthy neonates using wide-field digital imaging system (RetCam III) in a multi-center network in China leaded by Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine. The multi-center network will be built with the collaboration of eight hospitals from different parts of China.

DETAILED DESCRIPTION:
Studies reveal that ocular anomalies may also be found in healthy full-term babies. These abnormal ocular findings included subconjunctival haemorrhage, congenital microphthalmos, congenital corneal leukoma, posterior synechia, persistent pupillary membrane, congenital cataract, enlarged C/D ratio, retinal hamartoma versus retinoblastoma, optic nerve defects, macular pigment disorder and non-specific peripheral retinopathy. The highest proportion of these abnormal findings is retinal haemorrhages, accounting for 92% of abnormalities. Most retinal hemorrhages are benign and will finally self-resolve. However, sometimes it takes a long time for the hemorrhage to resolve. Some slow-resolving hemorrhages could obstruct the visual axis and may do great harm to visual development in critical period. Some neonatal eye diseases are time sensitive, such as retinoblastoma, and if found late, the best opportunity for effective treatment is missed, leading to irreversible visual impairment. Newborns are unable to express their discomforts or visual disorders as adults do and only through an examination, the neonatal eye diseases can be detected. Therefore, this screening protocol is designed to screen the otherwise healthy neonates in a multi-center network on neonatal ophthalmopathy and to achieve early diagnosis and timely treatment. All the neonates will undergo eye examination by using RetCam III. The external eye, pupillary light reflex, red reflex, opacity of refractive media, anterior chamber and posterior segments will be examined. The outcomes will be analyzed by a blinded specialist in order to discover serious congenital, hereditary and acquired diseases in the neonatal period of healthy newborns and to improve epidemiological information of neonatal ophthalmopathy. Neonatal ocular examination may play a positive role in promoting paediatric eye health to paediatricians and parents.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy neonates ( ≥37weeks' gestational age, weighing ≥2500 g, no evidence of systemic disease and an Apgar score of 7 or more.)

Exclusion Criteria:

* Preterm /Neonates with systemic diseases
* Neonates unable to undergo the examination

Ages: 2 Days to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Otherwise healthy neonates in a multicenter network in China
Sampling Method: Probability Sample
Enrollment: 30000 (Actual)
Dates: Start 2016-07; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
presence of ocular disease | 2 to 7 days after birth

CONTACTS AND LOCATIONS:
Overall Officials: Peiquan Zhao, MD, Principal Investigator — Xinhua Hospital, School of Medicine, Shanghai Jiaotong University, China
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided